CLINICAL TRIAL: NCT02831192
Title: International Multi-center Clinical Study on Microtransplantation for Treatment of Newly Diagnosed Elderly Acute Myeloid Leukemia (EAML)
Brief Title: Microtransplantation in Older Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EAML-MST
Record Dates: First submitted 2016-07-03; First posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MST（microtransplantation） (Experimental)
  Interventions: Biological: microtransplantation

INTERVENTIONS:
Biological: microtransplantation — HLA mismatched donor mobilized prepheral stem cell infusion

SUMMARY:
The purpose of this study is to see whether HLA-mismatched donor cells infusion with chemotherapy (microtransplantation，MST) could increase complete remission (CR) and improve survival in older patients with acute myeloid leukemia (AML)，the investigators conducted a prospective, multicenter clinical trial of HLA-mismatched MST to estimate outcomes and toxicities.

ELIGIBILITY:
Inclusion Criteria:

* de novo acute myeloid leukemia
* age 60-90
* have HLA mismatched donor

Exclusion Criteria:

* have no suitable donor or donor refused
* patient refused to accept donor cells

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Graft versus host disease | 1 month

SECONDARY OUTCOMES:
overall survival | 2 years
leukemia free survival | 2 years
complete remission rate | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: AI huisheng, MD, Study Chair — Affiliated Hospital of Academy of Military Medical Sciences
Locations (1):
- Affiliated Hospital of Academy of Military Medical Sciences ,, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided